CLINICAL TRIAL: NCT05576337
Title: Comparison of Neuromuscular Characteristics of Strict Vegetarians and Non-Vegetarians Women and Their Adaptations After 16 Weeks of Strength Training
Brief Title: Neuromuscular Characteristics of Strict Vegetarians and Non-Vegetarians Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Ronei Silveira Pinto, University Teacher/Doctor, Universidade Federal do Rio de Janeiro
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 52472821.6.0000.5347
Record Dates: First submitted 2022-09-23; First posted 2022-10-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hypertrophy
Keywords: Muscle mass; Muscle quality; Strength; Power
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict vegetarians (Experimental): Strict vegetarians women
  Interventions: Other: 16 weeks of strength training protocol
- non vegetarians (Experimental): Non vegetarians women
  Interventions: Other: 16 weeks of strength training protocol

INTERVENTIONS:
Other: 16 weeks of strength training protocol — 16 weeks of strength training protocol

SUMMARY:
A strict vegetarian diet includes only foods of plant-based origin and, despite being able to meet the nutritional needs of individuals of different ages, when correctly planned, it commonly offers a lower protein intake than a non-vegetarian diet. Daily protein intake directly influences the turnover of body proteins (synthesis vs. degradation rates), being important for the maintenance of skeletal muscle mass, tissue that performs metabolic functions in the body and enables the performance of tasks of daily living. In addition, the practice of strength training (ST) interferes in muscle mass increasing rates, also exerting an influence in muscle quality, strength and power increase, which are associated with better physical fitness, quality of life and health. To make these increases possible, especially in relation to morphological aspects, a higher protein intake than recommended for the general population is necessary (1.2 to 1.6 g/kg/day), which requires careful dietary planning, especially when the consumption of meat, eggs and dairy products, which are important sources of this nutrient, is excluded. Thus, the present study has two main objectives: to compare the neuromuscular characteristics of strict vegetarians (VE) and non-vegetarians (NV) (Phase 1 - cross-sectional) and the neuromuscular adaptations induced by 16 weeks of ST (Phase 2 - longitudinal).

DETAILED DESCRIPTION:
A strict vegetarian diet includes only foods of plant-based origin and, despite being able to meet the nutritional needs of individuals of different ages, when correctly planned, it commonly offers a lower protein intake than a non-vegetarian diet. Daily protein intake directly influences the turnover of body proteins (synthesis vs. degradation rates), being important for the maintenance of skeletal muscle mass, tissue that performs metabolic functions in the body and enables the performance of tasks of daily living. In addition, the practice of strength training (ST) interferes in muscle mass increasing rates, also exerting an influence in muscle quality, strength and power increase, which are associated with better physical fitness, quality of life and health. To make these increases possible, especially in relation to morphological aspects, a higher protein intake than recommended for the general population is necessary (1.2 to 1.6 g/kg/day), which requires careful dietary planning, especially when the consumption of meat, eggs and dairy products, which are important sources of this nutrient, is excluded. Thus, the present study has two main objectives: to compare the neuromuscular characteristics of strict vegetarians (VE) and non-vegetarians (NV) (Phase 1 - cross-sectional) and the neuromuscular adaptations induced by 16 weeks of ST (Phase 2 - longitudinal). For Phase 1, 140 healthy adults of both sexes (70 VE and 70 NV) will be recruited, who have been strength-untrained and who have adhered to the respective dietary pattern, both for at least 6 months. Participants will be instructed to perform the 3-day food record and count the number of steps for 5 days. Subsequently, they will undergo assessments of body composition, physical activity level and neuromuscular tests of the lower limbs (maximum strength, jumping power and muscle thickness of the quadriceps femoris, hamstring and gastrocnemius muscles). Comparisons of means between groups will be performed by the T test - independent. Results will be expressed as mean and standard deviation and the accepted significance level will be 5%. For Phase 2, 33 VE and 33 NV will be recruited (66 participants in total), who, in addition to meeting the eligibility criteria set out in Phase 1, are also available to participate in the strength training period. Participants will undergo the same assessments provided for in Phase 1 and must maintain their respective eating habits and patterns. At the 4th, 8th, 12th, and 16th weeks of ST, all participants will complete a new 3-day food record and perform step counts. In the 17th week, the initial evaluations will be repeated. Comparisons will be performed through two-way analysis of variance with repeated measures, considering the factors group (2 stratifications), time (2 stratifications) and group x time interaction. Results will be expressed as mean and standard deviation and the accepted significance level will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index until 30kg/m²
* Be a strict vegetarian or non-vegetarian for at least 6 months
* Not performing regular physical exercise for at least 6 months

Exclusion Criteria:

* Having chronic diseases, such as systemic arterial hypertension, diabetes mellitus, cardiomyopathy
* Present physical limitations or musculoskeletal problems, which contraindicate the performance of strength exercises
* Make use of a protein or amino acid food supplement, caffeine or other thermogenic substances

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Quadriceps femoris muscle thickness assessed by ultrasonography images | Change from baseline at 16 weeks of strength training
  Quadriceps femoris muscle thickness (vastus lateralis (VL) + rectus femoris (RF) + vastus medialis (VM) + vastus intermedius (VI) muscle thickness (MT, mm)) will be assessed by ultrasonography equipament. The RF and VI images will be assessed at two-thirds of the distance between the greater trochanter and the lateral epicondyle of the femur. VL images will be assessed at midpoint between greater trochanter and the lateal epicondyle of the femur. Thus, VM images will be assessed at the location corresponding to 30% of the distance between the lateral epicondyle and the greater trochanter of the femur. The images analisys will realized, posteriorly, by Image-J software.
Hamstrings muscle thickness assessed by ultrasonography images | Change from baseline at 16 weeks of strength training
  Hamstrings muscle thickness (i.e femural bíceps and semitendinosus muscle thickness; MT (mm)) will be assessed by ultrasonography images. Thi images will be obteined at 50% of distance between femur´s greater trochanter and the lateral line of the knee joint. In the image obtained, the muscle tissue between the adipose tissue interfaces will be identified, and the distance between these tissues will be defined as the muscle thickness. The analysis of the images will be carried out in the Image-J software.
Gastrocnemius muscle thickness assessed by ultrasonography images | Change from baseline at 16 weeks of strength training
  Will be asssesed by images obteined by ultrasonography equipament. The points for capturing the ultrasonography images of the gastrocnemius will be marked with a dermographic pen in the most medial cross-sectional area and with the greatest volume, verified with the probe. In the image obtained, the muscle tissue between the adipose tissue interfaces will be identified, and the distance between these tissues will be defined as the muscle thickness. The analysis of the images will be carried out in the Image-J software.

SECONDARY OUTCOMES:
Lower limb muscle power in the jumping performance test assessed by a contact mat | Change from baseline at 16 weeks of strength training
  To evaluate the muscle power of the lower limbs, a jump test with counter-movement bilaterally will be used. 3 to 5 submaximal jumps will be conducted for possible performance adjustments. At 5 minutes rest, the submaximal tests will be executed. The participant will perform the maximum jump as quickly and powerfully as possible, and the average of 3 jumps, separated by 30s, will be used as a performance result. The evaluations will be conducted on a contact mat which will automatically inform the performance of the participants
Rigth thigh dynamic muscle strength assessed by isokinetic dynamometer | Change from baseline at 16 weeks of strength training
  The right thigh muscle strength will be assessed using peak torque (PT, N.m) obteined by isokinetic dynamometer. Will be realized 5 maximal concentric isokinetic contractions of knee extension and flexion, with a velocity of 60º.s-1 and range of motion between zero (maximum extension) and 90º of knee flexion. In addition, will be realized 5 eccentric knee flexion contractions with the same speed and amplitude as in the previous test. Between each dynamic test, a 1-minute interval will be observed and, before performing each test, a submaximal familiarization series with the same number of repetitions, speed and range of motion will be performed. The participant will be instructed to perform all tests "as quickly and as hard as possible". In addition, the participant will receive verbal stimulation during the tests.
Knee extensors dynamic muscle strength assessed by one maximum repetition test | Change from baseline at 16 weeks of strength training
  Will be evaluated by 1 maximum repetition (1MR) test of knee extensors muscles to be performed in KONNEN GYM® equipments. The 1 maximum repetition test load (kg) will be estimated through trial and error. Lombardi correction coefficients will be used to adjust the load between trials. The exercise will consist of performing the concentric phase, starting from the initial position (90º of knee flexion) to the final phase (maximum knee extension), and returning to the initial position, eccentric phase. To minimize the effect of fatigue on the test result, 3-minute intervals will be observed for warm-up, as well as between each load increment. The 1MR load will be considered the one in which the participant can perform only one maximum repetition with cadence (2 seconds for the concentric phase and 2 seconds for the eccentric phase) and desired range of motion (from the position of 90º of knee flexion to the maximum knee extension position).
Knee flexors dynamic muscle strength assessed by one maximum repetition test | Change from baseline at 16 weeks of strength training
  Will be evaluated by 1 maximum repetition (1MR) test of hamstrings muscles to be performed in KONNEN GYM® flexion equipment. The 1 maximum repetition test load (kg) will be estimated through trial and error. Lombardi correction coefficients will be used to adjust the load between trials. The exercise will consist of performing the concentric phase, starting from the initial position (180º of knee extension) to the final phase (90° knee flexion), and returning to the initial position, eccentric phase. To minimize the effect of fatigue on the test result, 3-minute intervals will be observed for warm-up, as well as between each load increment. The 1MR load will be considered the one in which the participant can perform only one maximum repetition with cadence (2 seconds for the concentric phase and 2 seconds for the eccentric phase) and desired range of motion (from the position of 180º of knee extension to the 90° knee flexion position).
Plantar flexors dynamic muscle strength assessed by one maximum repetition test | Change from baseline at 16 weeks of strength training
  Will be evaluated by 1 maximum repetition (1MR) test of plantar flexors muscles to be performed in KONNEN GYM® plantar flexion equipment. The 1 maximum repetition test load (kg) will be estimated through trial and error. Lombardi correction coefficients will be used to adjust the load between trials. The exercise will consist of performing the concentric phase, starting from the initial position (45° of ankle flexion) to the final phase (45° ankle flexion), and returning to the initial position, eccentric phase. To minimize the effect of fatigue on the test result, 3-minute intervals will be observed for warm-up, as well as between each load increment. The 1MR load will be considered the one in which the participant can perform only one maximum repetition with cadence (2 seconds for the concentric phase and 2 seconds for the eccentric phase) and desired range of motion (from the position of 180º of knee extension to the 90° knee flexion position).
Quadriceps femoris muscle quality evaluated by echointensity through images obtained by ultrasonography. | Change from baseline at 16 weeks of strength training
  The muscle quality by echo-intensity of the quadriceps femoris muscle will be obtained from images collected for the measurement of muscle thickness, using an ultrasonography device. The largest muscle area of interest will be delimited without considering fascia and bone, and the analysis will be based on a gray scale histogram where 0 is black and 255 is white. The analysis will be performed using the same software (ImageJ, version 1.37, National Institutes of Health, USA) and the average of the values of three captured images will be used for further analysis.
Hamstrings muscle quality evaluated by echointensity through images obtained by ultrasonography. | Change from baseline at 16 weeks of strength training
  The muscle quality by echo-intensity of the hamstrings muscles will be obtained from images collected for the measurement of muscle thickness, using an ultrasonography device. The largest muscle area of interest will be delimited without considering fascia and bone, and the analysis will be based on a gray scale histogram where 0 is black and 255 is white. The analysis will be performed using the same software (ImageJ, version 1.37, National Institutes of Health, USA) and the average of the values of three captured images will be used for further analysis.
Gastrocnemius muscle quality evaluated by echointensity through images obtained by ultrasonography. | Change from baseline at 16 weeks of strength training in the gastrocnemius muscle quality evaluated by echointensity through images obtained by ultrasonography
  The muscle quality by echo-intensity of the gastrocnemius muscles will be obtained from images collected for the measurement of muscle thickness, using an ultrasonography device. The largest muscle area of interest will be delimited without considering fascia and bone, and the analysis will be based on a gray scale histogram where 0 is black and 255 is white. The analysis will be performed using the same software (ImageJ, version 1.37, National Institutes of Health, USA) and the average of the values of three captured images will be used for further analysis.
Right thigh muscle quality estimated by specific tension | Change from baseline at 16 weeks of strength training
  It will be determined by the ratio between the value of the concentric peak torque (N.m) of the right knee extensors and flexors, determined by an isokinetic dynamometer test, and the value of the lean mass (kg) of the right thigh, obtained by Dual Energy X-Ray Emission Absorptiometry, in which a region of interest of the thigh will be evaluated through the manual construction of a box.
Gastrocnemius muscle quality estimated by specific tension | Change from baseline at 16 weeks of strength training
  It will be determined by the ratio between the value of the one maximum repetition (Kg) of the right plantar flexors, determined by an one maximum repetition test, and the value of the lean mass (kg) of the right leg, obtained by Dual Energy X-Ray Emission Absorptiometry, in which a region of interest of the thigh will be evaluated through the manual construction of a box.
Daily protein intake relative to total body mass assessed by 3 day food record | At baseline, within 4, 8 and 12 weeks of starting strength training and with the end of the 16 weeks of strength training
  Daily protein intake relative to total body mass will be assessed by 3 day food record that will be realized by Dietbox software. The records must include the times, quantities in household measures and, when possible, the brand of the food product. In addition, each participant will make a photographic record of each meal (dish served/package/food), to assist in understanding food intake. A photographic material will be provided with the size of the portions to assist in filling in homemade measures. The records will be analyzed with the same software, preferably using the data registered in the Food Composition Table (TACO) (NEPA; UNICAMP, 2011), Food composition table: support for nutritional decision (PHILIPPI, 2016), Brazilian Table of Food Composition (TBCA) (USP; FORC, 2020) and food label.
Correlation between protein intake food and neuromuscular characteristics | Change from baseline at 16 weeks of strength training
  The protein food intake relative to total body mass assessed by 3 day food record will be correlated with neuromuscular characteristics (Quadriceps femoris, hamstrings and gastrocnemius muscle thickness assessed by ultrasonography images; lower limb muscle power in the jumping performance test assessed by a contact mat; rigth thigh dynamic muscle strength assessed by isokinetic dynamometer; knee extensors, knee flexors and plantar flexors dynamic muscle strength assessed by one maximum repetition test; quadriceps femoris, hamstrings and gastrocnemius muscle quality evaluated by echointensity through images obtained by ultrasonography; right thigh and gastrocnemius muscle quality estimated by specific tension).
Total food intake | At baseline, within 4, 8 and 12 weeks of starting strength training and with the end of the 16 weeks of strength training
  Total food intake will be assessed by 3 day food record ijn the same way that daily protein intake relative to total body mass outcome The total amounts (g, mg) of nutrients (calories, carbohydrates, fats, protein, amino acids, iron, zinc, calcium, selenium, vitamins D, B12) will be evaluated and relativized by body mass (proteins), ingested on the day and by snack.
Body composition assessed by Dual Energy X-Ray Emission Absorptiometry (DXA) | Change from baseline at 16 weeks of strength training
  The total and regional bone content (kg), boné mineral density (kg/cm²), fat (kg) and lean mass (kg) will be assessed with absorption by dual energy x-ray emission (DXA). During the test, participants will be positioned in supine position, aligned and centered on the examination table with hips and shoulders extended to initiate the X-ray scan. Also, they will be instructed to wear light clothes at the time of the assessment, which allow adequate body scanning, in addition to not wearing metal accessories. The radiation that the participant will be exposed during the evaluation is safe and less than 1μSv (BOLANOWSKI; NILSSON, 2001). The equipment will be calibrated before each scan according to the manufacturer's specifications. The obteined images will be evaluated later using the software (Encore versão 41.1, Lunar Prodgy Madison, USA).
Body composition assessed by anthropometry measurements | Change from baseline at 16 weeks of strength training
  The Body mass (kg) and Heigh (cm) will be assesed for the body mass index (BMI) calculation as inclusion criteria, that will be classified according world health organization (WHO, 2000) parameters. Participants will be evaluated wearing light clothes and barefoot on an ASIMED® scale with a resolution of 0.1 kg. The heigh will be assessed with wall scale. Perimeters (cm), skinfolds (mm), bone diameters and lengths (cm) also will be assessed. The total and regional body composition analisys will be realized. All measurements will follow the standardization protocol of measurements made by ISAK (International Society for the Advancement of Kinanthropometry) and will be assessed in the high side of the body, in duplicate, if necessary in triplicate, and the mean, mode or median will be used, as final result.
Physical activity level assessed by International Physical Activity Questionnaire | Change from baseline at 16 weeks of strength training
  Participants will receive a printed copy of the short version of the International Physical Activity Questionnaire, which is self-applied and validated for the Brazilian population (CRAIG et al., 2003; MATSUDO et al., 2001). The Questionnaires will be analyzed and classified according to the tool's categorical score as "low", "moderate" and "high" physical activity level.
Physical activity level assessed by daily step count | Change from baseline at 16 weeks of strength training
  The evaluation of the counting of the daily steps will be assessed by daily step count, that will be evaluated during 7 days at baseline and after 16s weeks of strength training. For this, participants will receive a pedometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ronei Silveira Pinto, Principal Investigator — Federal University of Rio Grande do Sul (UFRGS); Claúdia Dornelles Schneider, Study Director — Federal University of Healthy Sciences of Porto Alegre (UFCSPA)
Locations (1):
- Federal University of Rio Grande do Sul (UFRGS), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05576337/Prot_SAP_ICF_000.pdf